CLINICAL TRIAL: NCT02679703
Title: Polarity Action in Electrical Stimulation Transcutaneous for Treatment of Graft Donor Areas in Patients Autogenous Burned: Blind Randomized Clinical Trial
Brief Title: Polarity Action in Electrical Stimulation Transcutaneous Donors for Treatment Areas Burned Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Elaine Caldeira de Oliveira Guirro, Principal Investigator, University of Sao Paulo
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 8639
Record Dates: First submitted 2016-02-06; First posted 2016-02-10 (Estimated); Last update posted 2016-02-10 (Estimated); Status verified 2016-02

CONDITIONS: Burn
MeSH Terms: conditions — Burns | interventions — Transcutaneous Electric Nerve Stimulation; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- High voltage (Experimental): The applied parameters of high voltage electrical stimulation are medium voltage of 100 volts, an increase in the course of the session, frequency of 10 Hz, with application in the donor areas of thigh or scalp for 40 minutes, 25% above of level engine daily until complete epithelialization, and removal of the dressing type rayon.
  Interventions: Device: High voltage
- Neuromuscular transcutaneous electrical stimulation (TENS) (Experimental): 10 Hz, 40 min, 200 μs and 25% above of motor level
  Interventions: Device: Neuromuscular transcutaneous electrical stimulation (TENS)
- Control Group (Experimental): There will be no intervention
  Interventions: Other: Control Group

INTERVENTIONS:
Device: High voltage — Electrical stimulation treatments will be made in donor areas (scalp and thigh) in patients burns
  Arms: High voltage
Device: Neuromuscular transcutaneous electrical stimulation (TENS) — Electrical stimulation treatments will be made in donor areas (scalp and thigh) in patients burns.
  Arms: Neuromuscular transcutaneous electrical stimulation (TENS)
Other: Control Group — The control group will not have electrical stimulation however, will be evaluated with digital digital imaging, thermography imaging, skin hardness and subjective pain and healing scales
  Arms: Control Group

SUMMARY:
To evaluate the effect of the polarity of the electric current in healing.

DETAILED DESCRIPTION:
The objective of this study is to evaluate the effect of the polarity of the current in healing. Both will be compared to the effects of electrical stimulation of high voltage (HVES) and neuromuscular transcutaneous electrical stimulation (TENS) in the treatment of donor sites (DA) of burn patients. It is a prospective, controlled clinical, randomized, blinded. Will be assessed 60 subjects aged 18-59 years, of both sexes, underwent the surgical procedure of grafting (PCE) were randomly divided into small blocks 5:5:5 three groups: undergoing therapeutic procedure with HVES undergoing therapeutic procedure with TENS and control. Therapeutic procedures will be applied around the DA, thigh or scalp, after 24 hours of PCE until complete healing. The variables will be the healing time estimated by the removal of the dressing rayon, clinical evaluation, scar quality, the Vancouver scale; pain, the pain numerical scale evaluation (PNS); blood perfusion by thermography; quality of healing by digital imaging, quantification of areas of crusts by the software Image J; skin biomechanical aspects as firmness, the durometer being performed reassessment at the end of treatment. Data will be submitted to analysis of normality by the Shapiro-Wilk test and the effect of behavior among groups and pre- and post-intervention will be evaluated by ANOVA-two way followed by post-hoc (Bonferroni) or Friedman, with p <0.05. Comparing groups, before a normal distribution is applied ANOVA followed by Tukey, and otherwise will be applied the Kruskal-Wallis test and post-hoc Dunn, p<0.05.

ELIGIBILITY:
Inclusion Criteria:

* Victims of second deep degree and third degree burns, aged between 18 and 59 years
* Both sexes
* Underwent the surgical procedure of grafting (PCE) with donor area of the scalp or thigh thick standardized mean (0.20 mm).

Exclusion Criteria:

* Diabetes,
* Infectious processes
* Use of medications that alter the healing process (corticosteroids, chemotherapy, radiotherapy, among others)
* Cognitive impairment
* Agreeing not to sign the Consent Form and Clarified or that do not fit the inclusion criteria described.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2016-02; Primary Completion 2016-02 (Actual); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Time | One year
  We will count the time it takes days to remove the dressing rayon in donor areas.

SECONDARY OUTCOMES:
Numerical Pain Scale | One year
  we will evaluate the patient's pain before and after application of electro stimulation

IPD SHARING:
Plan to Share IPD: Undecided